CLINICAL TRIAL: NCT06226805
Title: A Multicenter, Double-blinded, Placebo-controlled, Single Ascending Dose, Two-part, Randomized, Phase 2 Clinical Trial to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BB-031 in Acute Ischemic Stroke Patients
Brief Title: Study of BB-031 in Acute Ischemic Stroke Patients (RAISE)
Acronym: RAISE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Basking Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BB-031-CLIN-201
Record Dates: First submitted 2024-01-07; First posted 2024-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Wake-up stroke; Large vessel occlusion; Intracranial hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Stroke; Intracranial Hemorrhages | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will receive a single dose of blinded investigational drug or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BB-031 (Experimental): A single dose of BB-031 will be administered via IV bolus injection
  Interventions: Drug: BB-031
- Placebo (Placebo Comparator): A single dose of matching placebo will be administered via IV bolus injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BB-031 — Solution for injection
  Other Names: DTRI-031
  Arms: BB-031
Drug: Placebo — 0.9% sodium chloride for injection
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ascending doses (Part A) and selected doses (Part B) of BB-031 in acute ischemic stroke patients presenting within 24 hours of stroke onset.

Participants will be randomized to receive one dose of either the investigational drug or placebo and will be followed for 90 days. A total of 228 patients are planned in this study.

DETAILED DESCRIPTION:
This is a two-part, randomized, placebo-controlled, double-blinded study in acute ischemic stroke patients. In Part A, up to 48 participants will be randomized in a 3:1 ratio (investigational drug: placebo) into 1 of 3 planned ascending dose groups to determine the dose levels to be studied in Part B. Two dose levels will be chosen based upon a review of all available data including safety, PK, PD and preliminary efficacy. In Part B, approximately 180 participants will be randomized to receive a single dose of two sequential dose levels of study drug or placebo.

All participants will be screened for participation after confirmed diagnosis of an anterior circulation ischemic stroke by neurovascular imaging. Enrolled participants will be followed for 90 days. Radiological outcomes will be assessed by a central blinded reviewer. A Data Safety Monitoring Committee will review safety and preliminary efficacy data throughout the study as outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke
* 18 years or older
* Anterior circulation intra-cranial occlusion
* NIHSS score >3
* Onset of stroke symptoms within 24 hours of enrollment

Exclusion Criteria:

* Large volume ischemic stroke
* Intracranial hemorrhage on baseline imaging or previous intracranial hemorrhage
* Chronic intracranial occlusion
* Weight >125kg
* Administration of thrombolytic drug or glycoprotein IIb/IIIa inhibitors
* Ongoing clinically significant coagulopathy, history of bleeding disorder or other conditions for high-risk bleeding or active uncontrolled bleeding
* Prior stroke within 90 days
* Unable to undergo a contrast brain perfusion scan with either MRI or CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Symptomatic Intracranial Hemorrhage (sICH) | 24 hours
  Proportion of participants having a sICH

SECONDARY OUTCOMES:
Asymptomatic intracranial hemorrhage (non-symptomatic-ICH) | 24 hours
  Proportion of participants having a non-symptomatic-ICH
Adverse Events (AEs) | 24 hours
  Incidence and severity of treatment-emergent AEs

OTHER OUTCOMES:
Mortality | 30 days, 90 days
  All-cause mortality
Pharmacokinetic (PK) Plasma Level Assessment | 48 hours
  Plasma levels of study drug
Pharmacokinetic (PK) Parameter | 48 hours
  Cmax
Pharmacodynamic (PD) Assessment | 72 hours
  Level of free circulating von Willibrand Factor
Pharmacodynamic (PD) Assessment | 72 hours
  von Willibrand Factor activity
Recanalization | 2-9 hours
  Proportion of participants with recanalization
Endovascular Thrombectomy (EVT) | 6 hours
  Proportion of participants where EVT was not performed due to clinical improvement or evidence of recanalization
Stroke lesion volume | 24 hours
  Assessed by MRI or CT
National Institutes of Health Stroke Scale (NIHSS) Score | 24 hours, 48 hours, hospital discharge and Day 90
  Change from baseline score (total score 0 to 42, with 0 representing no abnormality
Modified Rankin Scale (mRS) Score | Day 90
  Change from baseline score, where 0=no symptoms and 6=dead
ICU length of stay | Up to Day 90
  Duration of ICU stay
Hospitalization length of stay | Up to Day 90
  Duration of hospitalization
Successful reperfusion after first pass EVT | 6 hours
  Proportion of subjects with successful reperfusion after first pass EVT

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Hill, MD, Principal Investigator — University of Calgary; Shahid M Nimjee, MD, PhD, Principal Investigator — Ohio State University
Locations (23):
- United States (14):
  - HonorHealth Bob Bove Neuroscience Institute, Scottsdale, Arizona
  - Mills Peninsula Medical Center, Burlingame, California
  - MemorialCare Long Beach Medical Center, Long Beach, California
  - California Pacific Medical Center, San Francisco, California
  - Pacific Neurosciences Institute at Saint John's Physician Partners, Torrance, California
  - Baptist Health Medical Center, Jacksonville, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - WakeMed, Raleigh, North Carolina
  - The Ohio State University, Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Valley Baptist Medical Center - Harlingen, Harlingen, Texas
  - Memorial Hermann Hospital, Houston, Texas
- Australia (6):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No